CLINICAL TRIAL: NCT03100656
Title: Solving EPHX2 and Polyunsaturated Fatty Acid Interactions in Anorexia Nervosa
Brief Title: Study of Food Aversion in Patients With Anorexia Nervosa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Toronto (Other); University of California, Davis (Other)
Responsible Party: Principal Investigator, Pei-an (Betty) Shih, Associate Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R01MH106781 (NIH)
Record Dates: First submitted 2017-03-03; First posted 2017-04-04 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Anorexia Nervosa
Keywords: psychopathology; treatment; epoxide hydrolases; polyunsaturated fatty acids; eicosanoids
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anorexia nervosa I (Other): Anorexia nervosa with BMI <=17.5 kg/m² or BMI >17.5 kg/m² with regular binge-purge episodes
  Interventions: Other: A breakfast sandwich
- Anorexia nervosa II (Other): Anorexia nervosa with BMI > 18.5 kg/m² for at least 12 months.
  Interventions: Other: A breakfast sandwich
- Controls (Other): Healthy control women
  Interventions: Other: A breakfast sandwich

INTERVENTIONS:
Other: A breakfast sandwich — A meat-based breakfast sandwich

SUMMARY:
This study uses a meal-challenge protocol to assess if patients with anorexia nervosa show a differential metabolism in response to food in comparison to healthy controls. This study determines how heritable and biochemical factors influence food metabolism in anorexia nervosa in order to develop more effective treatment strategies.

DETAILED DESCRIPTION:
Anorexia nervosa is a brain-based disorder that often leads to serious health consequences including death. The EPHX2 gene has been identified as a susceptibility gene for anorexia nervosa. This study utilizes a multi-omics biomarker system approach to investigate how genetic factors interact with dietary factors to influence food aversion, psychopathology, and clinical outcome in patients with anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Ill AN subjects will meet current Diagnostic and Statistical Manual of Mental Disorders (DSM V) diagnosis of AN, body mass index (BMI) between 11 kg/m² and 17.5 kg/m², or BMI > 17.5 kg/m² with active eating disorder symptoms.
* Recovered AN must meet the following criteria at time of study entry: 1) Current or past DSM V diagnosis of AN; 2) BMI between 18.5 kg/m2 and 30 kg/m2; 3) Having maintained a BMI of >18.5 for at least one year.
* Control must be healthy adolescent or woman negative on our screen for AN, other Axis I psychiatric illnesses, and having maintained a BMI of between 18.5-30 kg/m² since the age of 18.

Exclusion Criteria:

* Exclusion criteria for AN and control subjects include: Organic brain syndrome, schizophrenia and schizoaffective disorder, untreated thyroid disease, renal disease, hepatic disease, and the regular use of fish-oil containing supplements within the last three months of the study. All pregnant and lactating individuals will be excluded.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-11-10 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of metabolism biomarker | 2 hours
  Percentage change of metabolism marker
Food aversion/anxiety | 2 hours
  Percentage change of food aversion/anxiety score

SECONDARY OUTCOMES:
Weight | 6 and 12 months
  Change in body weight, kg
Psychopathology | 6 and 12 months
  Percentage change in eating disorder psychopathology score

CONTACTS AND LOCATIONS:
Overall Officials: Pei-an (Betty) Shih, MPM, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- UC San Diego Altman Clinical and Translational Research Institute, La Jolla, California, United States
- Program for Eating Disorders, Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shih PB. Integrating multi-omics biomarkers and postprandial metabolism to develop personalized treatment for anorexia nervosa. Prostaglandins Other Lipid Mediat. 2017 Sep;132:69-76. doi: 10.1016/j.prostaglandins.2017.02.002. Epub 2017 Feb 21. PMID 28232135
- [Background] Shih PA, Woodside DB. Contemporary views on the genetics of anorexia nervosa. Eur Neuropsychopharmacol. 2016 Apr;26(4):663-73. doi: 10.1016/j.euroneuro.2016.02.008. Epub 2016 Feb 20. PMID 26944296
- [Background] Shih PB, Yang J, Morisseau C, German JB, Zeeland AA, Armando AM, Quehenberger O, Bergen AW, Magistretti P, Berrettini W, Halmi KA, Schork N, Hammock BD, Kaye W. Dysregulation of soluble epoxide hydrolase and lipidomic profiles in anorexia nervosa. Mol Psychiatry. 2016 Apr;21(4):537-46. doi: 10.1038/mp.2015.26. Epub 2015 Mar 31. PMID 25824304
- [Result] Nguyen N, Dow M, Woodside B, German JB, Quehenberger O, Shih PB. Food-Intake Normalization of Dysregulated Fatty Acids in Women with Anorexia Nervosa. Nutrients. 2019 Sep 13;11(9):2208. doi: 10.3390/nu11092208. PMID 31540208
- See also: Food Aversion Study For Anorexia Nervosa at University of California, San Diego — https://g3garcia.wixsite.com/eatdisordersresearch